CLINICAL TRIAL: NCT04145414
Title: Cerebrospinal Fluid Movements Through Interventricular Foramina in Phase Contrast Magnetic Resonance Imaging (PC-MRI)
Acronym: MLCSFIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2019/425
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: CSF Circulation Disorder; Foramen; Monro, Obstruction; Mri
Keywords: CSF; PC-MRI; interventricular foramina
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral magnetic resonance imaging x2 (Experimental): Cerebral MRI performed at enrolment visit and at +6 weeks (maximum)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Reproductibility test assessed with MRI for cerebrospinal fluid movements

SUMMARY:
Assess the reproductibility of PC-MRI for cerebrospinal fluid movements through the interventricular foramina on volunteer subjects.

DETAILED DESCRIPTION:
It is a monocentric interventional prospective study. Each subject will have to pass two MRI. Phase contrast MRI (PC-MRI) will be calibrated for each subject by assessing the optimal encoding velocity. Three sequences including the aqueduct and the two interventricular foramina (IVF) will be done. The signal will be analysed by syngo.via software after defining by two different investigators the region of interest (ROI) which correspond to the IVF or the aqueductal lumen. Descriptive statistics will test the intra-individual and inter-observer consistency based on 4 flow parameters.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination score > 28/30

Exclusion Criteria:

* MRI contraindication
* Medical or surgical history related to following pathologies: nervous system disease, cardiac arrhythmia, cardiac or respiratory insufficiency.
* Long-term medical treatment
* Ongoing pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
PC-MRI procedure reproductibility | week 6
  Test-retest reproducibility of double measures (2nd measure at +48 hours minimum +6 weeks maximum) of 4 cerebrospinal liquid (CSL) flow parameters during PC-MRI.
  CSL flow through interventricular foramina will be measured within healthy volunteers, and 4 intraclass correlation coefficients (ICC) will be calculated.
  The test-retest coefficient will be considered satisfactory if > or = to 0.75 .

CONTACTS AND LOCATIONS:
Overall Officials: Laurent TATU, MD, PhD, Principal Investigator — CHU Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No